CLINICAL TRIAL: NCT02328885
Title: Prophylactic Infusion of Donor Lymphocytes in Cord Blood Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Banc de Sang i Teixits (Other)
Collaborators: Hospital Vall d'Hebron (Other); Hospital de Sant Pau (Other); Hospital Universitari de Bellvitge (Other); Germans Trias i Pujol Hospital (Other); Fundacion IMIM (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I.2013.004
Record Dates: First submitted 2014-12-16; First posted 2014-12-31 (Estimated); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Leukemia
Keywords: high-risk acute leukemia; graft versus leukemia; DLI; UCBT
MeSH Terms: conditions — Leukemia

STUDY DESIGN:
Intervention Model Description: DLI
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): DLI of the 20 fraction of the UCBT
  Interventions: Drug: DLI of the 20 fraction of the UCBT

INTERVENTIONS:
Drug: DLI of the 20 fraction of the UCBT — Administration of 20 fraction of the UCBT

SUMMARY:
Pilot, multicentric, open-label, single-arm, phase I-II clinical trial to evaluate the safety and efficacy of a novel Umbilical Cord Blood Transplantation (UCBT) platform, that consists of a UCBT of the 80 fraction, followed by a Donor Lymphocyte Infusion (DLI) of the 20 fraction (between 60 and 90 days after transplantation).

DETAILED DESCRIPTION:
Multicenter, open-label, single-arm, phase I-II pilot study in which a minimum of 20 patients will enter the study with the primary objective to assess the safety and secondary objective to assess efficacy in relation to immune reconstitution followed by a new platform of treatment consisting of initial cord blood unit 80 fraction transplantation, followed by a prophylactic donor lymphocyte infusion (DLI) of the fraction 20 of the cord blood unit. The second infusion will take place between 60 and 90 days after transplantation.

ELIGIBILITY:
Inclusion Criteria:

At the time of transplantation:

* Patients under 60 years with proposal UCBT according to assistance protocol
* Diagnosis of high-risk acute leukemia with an indication of allogenic transplantation
* Frozen UCB bag split into two bags: one with the 80% of the product and another with the 20%
* Presence of at least 1.2E9 total nucleated cells and> 1E5 CD34 / kg and> 6E6 CD34 + in fraction 80%
* 4/6 or better compatibility taking Human Leukocyte Antigen (HLA) HLA-A, HLA-B by antigenic resolution and DRB1 by allelic resolution
* The patient (or legal representative if required) has signed the informed consent

At the time of DLI:

* Documented cord blood engraftment
* The patient has had no Graft Versus Host Disease (GVHD) during the first 60 days post-transplantation or, if present, receives less than 10 milligrams of prednisone at the time of the DLI or <0.2 mg / kg / day of prednisone for pediatric patients (<16 years).
* The patient has less than 200 CD4 + cells per microliter on peripheral blood at 60 days (± 7 days) post-transplantation
* The patient (or legal representative if required) has signed the informed consent

Exclusion Criteria:

At the time of transplantation:

* Simultaneous participation in another clinical trial or treatment with other research phase product within 30 days prior to inclusion in the study.
* Pregnant women or those who intend to become pregnant within 12 months after the signing of the informed consent or not taking proper contraceptive measures according to investigator criteria.
* Breastfeeding women
* Other pathologies or circumstances that may compromise the patient's participation in the study according to the criteria of the investigator.

At the time of DLI:

* Grade III-IV GVHD after allogeneic UCB
* Prednisone treatment (> 10 mg total per day in adults or> 0.2 mg / kg / day prednisone for pediatric patients)

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Safety assessment | 1 year
  Adverse events

SECONDARY OUTCOMES:
Immune reconstitution: | 1 year
  Subpopulations of Lymphocytes T: CD4 and CD8
Immunological reconstitution: | 1 year
  NK cells
Immune regeneration | 1 year
  Lymphocytes B
Infections in treated patients | 1 year
  Incidence of infections
Infections in the treated patients | 1 year
  Type of infections
Relapse of leukemia | 1 year
  Incidence of relapse
Survival curves | 1 year
  Global and disease-free survival
Mortality | 1 year
  Incidence of early and late mortality

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Querol, PhD, Principal Investigator — Banc de Sang i Teixits
Locations (4):
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital de Sant Pau, Barcelona
  - Hospital Vall Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dohner H, Estey EH, Amadori S, Appelbaum FR, Buchner T, Burnett AK, Dombret H, Fenaux P, Grimwade D, Larson RA, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz MA, Sierra J, Tallman MS, Lowenberg B, Bloomfield CD; European LeukemiaNet. Diagnosis and management of acute myeloid leukemia in adults: recommendations from an international expert panel, on behalf of the European LeukemiaNet. Blood. 2010 Jan 21;115(3):453-74. doi: 10.1182/blood-2009-07-235358. Epub 2009 Oct 30. PMID 19880497
- [Background] Cornelissen JJ, van Putten WL, Verdonck LF, Theobald M, Jacky E, Daenen SM, van Marwijk Kooy M, Wijermans P, Schouten H, Huijgens PC, van der Lelie H, Fey M, Ferrant A, Maertens J, Gratwohl A, Lowenberg B. Results of a HOVON/SAKK donor versus no-donor analysis of myeloablative HLA-identical sibling stem cell transplantation in first remission acute myeloid leukemia in young and middle-aged adults: benefits for whom? Blood. 2007 May 1;109(9):3658-66. doi: 10.1182/blood-2006-06-025627. Epub 2007 Jan 9. PMID 17213292
- [Background] Koreth J, Schlenk R, Kopecky KJ, Honda S, Sierra J, Djulbegovic BJ, Wadleigh M, DeAngelo DJ, Stone RM, Sakamaki H, Appelbaum FR, Dohner H, Antin JH, Soiffer RJ, Cutler C. Allogeneic stem cell transplantation for acute myeloid leukemia in first complete remission: systematic review and meta-analysis of prospective clinical trials. JAMA. 2009 Jun 10;301(22):2349-61. doi: 10.1001/jama.2009.813. PMID 19509382
- [Background] Lodewyck T, Cornelissen JJ. Allogeneic stem cell transplantation in acute myeloid leukemia: a risk-adapted approach. Blood Rev. 2008 Nov;22(6):293-302. doi: 10.1016/j.blre.2008.03.008. Epub 2008 May 1. PMID 18455284
- [Background] Messner HA. How good is allogeneic transplantation for high-risk patients with AML? Best Pract Res Clin Haematol. 2006;19(2):329-32. doi: 10.1016/j.beha.2005.11.007. PMID 16516130
- [Background] Schlenk RF, Dohner K, Mack S, Stoppel M, Kiraly F, Gotze K, Hartmann F, Horst HA, Koller E, Petzer A, Grimminger W, Kobbe G, Glasmacher A, Salwender H, Kirchen H, Haase D, Kremers S, Matzdorff A, Benner A, Dohner H. Prospective evaluation of allogeneic hematopoietic stem-cell transplantation from matched related and matched unrelated donors in younger adults with high-risk acute myeloid leukemia: German-Austrian trial AMLHD98A. J Clin Oncol. 2010 Oct 20;28(30):4642-8. doi: 10.1200/JCO.2010.28.6856. Epub 2010 Aug 30. PMID 20805454
- [Background] Appelbaum FR. Pursuing the goal of a donor for everyone in need. N Engl J Med. 2012 Oct 18;367(16):1555-6. doi: 10.1056/NEJMe1209982. No abstract available. PMID 23075182
- [Background] Barker JN, Byam CE, Kernan NA, Lee SS, Hawke RM, Doshi KA, Wells DS, Heller G, Papadopoulos EB, Scaradavou A, Young JW, van den Brink MR. Availability of cord blood extends allogeneic hematopoietic stem cell transplant access to racial and ethnic minorities. Biol Blood Marrow Transplant. 2010 Nov;16(11):1541-8. doi: 10.1016/j.bbmt.2010.08.011. Epub 2010 Aug 25. PMID 20800103
- [Background] Byrd JC, Mrozek K, Dodge RK, Carroll AJ, Edwards CG, Arthur DC, Pettenati MJ, Patil SR, Rao KW, Watson MS, Koduru PR, Moore JO, Stone RM, Mayer RJ, Feldman EJ, Davey FR, Schiffer CA, Larson RA, Bloomfield CD; Cancer and Leukemia Group B (CALGB 8461). Pretreatment cytogenetic abnormalities are predictive of induction success, cumulative incidence of relapse, and overall survival in adult patients with de novo acute myeloid leukemia: results from Cancer and Leukemia Group B (CALGB 8461). Blood. 2002 Dec 15;100(13):4325-36. doi: 10.1182/blood-2002-03-0772. Epub 2002 Aug 1. PMID 12393746
- [Background] Schlenk RF, Dohner K, Krauter J, Frohling S, Corbacioglu A, Bullinger L, Habdank M, Spath D, Morgan M, Benner A, Schlegelberger B, Heil G, Ganser A, Dohner H; German-Austrian Acute Myeloid Leukemia Study Group. Mutations and treatment outcome in cytogenetically normal acute myeloid leukemia. N Engl J Med. 2008 May 1;358(18):1909-18. doi: 10.1056/NEJMoa074306. PMID 18450602
- [Background] Krauter J, Wagner K, Schafer I, Marschalek R, Meyer C, Heil G, Schaich M, Ehninger G, Niederwieser D, Krahl R, Buchner T, Sauerland C, Schlegelberger B, Dohner K, Dohner H, Schlenk RF, Ganser A. Prognostic factors in adult patients up to 60 years old with acute myeloid leukemia and translocations of chromosome band 11q23: individual patient data-based meta-analysis of the German Acute Myeloid Leukemia Intergroup. J Clin Oncol. 2009 Jun 20;27(18):3000-6. doi: 10.1200/JCO.2008.16.7981. Epub 2009 Apr 20. PMID 19380453
- [Background] MATHE G, AMIEL JL, SCHWARZENBERG L, CATTAN A, SCHNEIDER M, DEVRIES MJ, TUBIANA M, LALANNE C, BINET JL, PAPIERNIK M, SEMAN G, MATSUKURA M, MERY AM, SCHWARZMANN V, FLAISLER A. SUCCESSFUL ALLOGENIC BONE MARROW TRANSPLANTATION IN MAN: CHIMERISM, INDUCED SPECIFIC TOLERANCE AND POSSIBLE ANTI-LEUKEMIC EFFECTS. Blood. 1965 Feb;25:179-96. No abstract available. PMID 14267694
- [Background] Horowitz MM, Gale RP, Sondel PM, Goldman JM, Kersey J, Kolb HJ, Rimm AA, Ringden O, Rozman C, Speck B, et al. Graft-versus-leukemia reactions after bone marrow transplantation. Blood. 1990 Feb 1;75(3):555-62. PMID 2297567
- [Background] Zittoun RA, Mandelli F, Willemze R, de Witte T, Labar B, Resegotti L, Leoni F, Damasio E, Visani G, Papa G, et al. Autologous or allogeneic bone marrow transplantation compared with intensive chemotherapy in acute myelogenous leukemia. European Organization for Research and Treatment of Cancer (EORTC) and the Gruppo Italiano Malattie Ematologiche Maligne dell'Adulto (GIMEMA) Leukemia Cooperative Groups. N Engl J Med. 1995 Jan 26;332(4):217-23. doi: 10.1056/NEJM199501263320403. PMID 7808487
- [Background] Cassileth PA, Harrington DP, Appelbaum FR, Lazarus HM, Rowe JM, Paietta E, Willman C, Hurd DD, Bennett JM, Blume KG, Head DR, Wiernik PH. Chemotherapy compared with autologous or allogeneic bone marrow transplantation in the management of acute myeloid leukemia in first remission. N Engl J Med. 1998 Dec 3;339(23):1649-56. doi: 10.1056/NEJM199812033392301. PMID 9834301
- [Background] Arora M, Nagaraj S, Wagner JE, Barker JN, Brunstein CG, Burns LJ, Defor TE, McMillan ML, Miller JS, Weisdorf DJ. Chronic graft-versus-host disease (cGVHD) following unrelated donor hematopoietic stem cell transplantation (HSCT): higher response rate in recipients of unrelated donor (URD) umbilical cord blood (UCB). Biol Blood Marrow Transplant. 2007 Oct;13(10):1145-52. doi: 10.1016/j.bbmt.2007.06.004. Epub 2007 Jul 27. PMID 17889350
- [Background] Laughlin MJ, Eapen M, Rubinstein P, Wagner JE, Zhang MJ, Champlin RE, Stevens C, Barker JN, Gale RP, Lazarus HM, Marks DI, van Rood JJ, Scaradavou A, Horowitz MM. Outcomes after transplantation of cord blood or bone marrow from unrelated donors in adults with leukemia. N Engl J Med. 2004 Nov 25;351(22):2265-75. doi: 10.1056/NEJMoa041276. PMID 15564543
- [Background] Barker JN, Davies SM, DeFor T, Ramsay NK, Weisdorf DJ, Wagner JE. Survival after transplantation of unrelated donor umbilical cord blood is comparable to that of human leukocyte antigen-matched unrelated donor bone marrow: results of a matched-pair analysis. Blood. 2001 May 15;97(10):2957-61. doi: 10.1182/blood.v97.10.2957. PMID 11342417
- [Background] Atsuta Y, Suzuki R, Nagamura-Inoue T, Taniguchi S, Takahashi S, Kai S, Sakamaki H, Kouzai Y, Kasai M, Fukuda T, Azuma H, Takanashi M, Okamoto S, Tsuchida M, Kawa K, Morishima Y, Kodera Y, Kato S; Japan Cord Blood Bank Network. Disease-specific analyses of unrelated cord blood transplantation compared with unrelated bone marrow transplantation in adult patients with acute leukemia. Blood. 2009 Feb 19;113(8):1631-8. doi: 10.1182/blood-2008-03-147041. Epub 2008 Dec 22. PMID 19104080
- [Background] Eapen M, Rubinstein P, Zhang MJ, Stevens C, Kurtzberg J, Scaradavou A, Loberiza FR, Champlin RE, Klein JP, Horowitz MM, Wagner JE. Outcomes of transplantation of unrelated donor umbilical cord blood and bone marrow in children with acute leukaemia: a comparison study. Lancet. 2007 Jun 9;369(9577):1947-54. doi: 10.1016/S0140-6736(07)60915-5. PMID 17560447
- [Background] Hwang WY, Samuel M, Tan D, Koh LP, Lim W, Linn YC. A meta-analysis of unrelated donor umbilical cord blood transplantation versus unrelated donor bone marrow transplantation in adult and pediatric patients. Biol Blood Marrow Transplant. 2007 Apr;13(4):444-53. doi: 10.1016/j.bbmt.2006.11.005. Epub 2007 Feb 15. PMID 17382250
- [Background] Takahashi S, Ooi J, Tomonari A, Konuma T, Tsukada N, Oiwa-Monna M, Fukuno K, Uchiyama M, Takasugi K, Iseki T, Tojo A, Yamaguchi T, Asano S. Comparative single-institute analysis of cord blood transplantation from unrelated donors with bone marrow or peripheral blood stem-cell transplants from related donors in adult patients with hematologic malignancies after myeloablative conditioning regimen. Blood. 2007 Feb 1;109(3):1322-30. doi: 10.1182/blood-2006-04-020172. Epub 2006 Oct 12. PMID 17038536
- [Background] Kumar P, Defor TE, Brunstein C, Barker JN, Wagner JE, Weisdorf DJ, Burns LJ. Allogeneic hematopoietic stem cell transplantation in adult acute lymphocytic leukemia: impact of donor source on survival. Biol Blood Marrow Transplant. 2008 Dec;14(12):1394-400. doi: 10.1016/j.bbmt.2008.09.021. PMID 19041062
- [Background] Rocha V, Labopin M, Sanz G, Arcese W, Schwerdtfeger R, Bosi A, Jacobsen N, Ruutu T, de Lima M, Finke J, Frassoni F, Gluckman E; Acute Leukemia Working Party of European Blood and Marrow Transplant Group; Eurocord-Netcord Registry. Transplants of umbilical-cord blood or bone marrow from unrelated donors in adults with acute leukemia. N Engl J Med. 2004 Nov 25;351(22):2276-85. doi: 10.1056/NEJMoa041469. PMID 15564544
- [Background] Verneris MR, Brunstein CG, Barker J, MacMillan ML, DeFor T, McKenna DH, Burke MJ, Blazar BR, Miller JS, McGlave PB, Weisdorf DJ, Wagner JE. Relapse risk after umbilical cord blood transplantation: enhanced graft-versus-leukemia effect in recipients of 2 units. Blood. 2009 Nov 5;114(19):4293-9. doi: 10.1182/blood-2009-05-220525. Epub 2009 Aug 25. PMID 19706886
- [Background] Rodrigues CA, Sanz G, Brunstein CG, Sanz J, Wagner JE, Renaud M, de Lima M, Cairo MS, Furst S, Rio B, Dalley C, Carreras E, Harousseau JL, Mohty M, Taveira D, Dreger P, Sureda A, Gluckman E, Rocha V. Analysis of risk factors for outcomes after unrelated cord blood transplantation in adults with lymphoid malignancies: a study by the Eurocord-Netcord and lymphoma working party of the European group for blood and marrow transplantation. J Clin Oncol. 2009 Jan 10;27(2):256-63. doi: 10.1200/JCO.2007.15.8865. Epub 2008 Dec 8. PMID 19064984
- [Background] Gutman JA, Leisenring W, Appelbaum FR, Woolfrey AE, Delaney C. Low relapse without excessive transplant-related mortality following myeloablative cord blood transplantation for acute leukemia in complete remission: a matched cohort analysis. Biol Blood Marrow Transplant. 2009 Sep;15(9):1122-9. doi: 10.1016/j.bbmt.2009.05.014. PMID 19660726
- [Background] Ruggeri L, Capanni M, Urbani E, Perruccio K, Shlomchik WD, Tosti A, Posati S, Rogaia D, Frassoni F, Aversa F, Martelli MF, Velardi A. Effectiveness of donor natural killer cell alloreactivity in mismatched hematopoietic transplants. Science. 2002 Mar 15;295(5562):2097-100. doi: 10.1126/science.1068440. PMID 11896281
- [Background] Willemze R, Rodrigues CA, Labopin M, Sanz G, Michel G, Socie G, Rio B, Sirvent A, Renaud M, Madero L, Mohty M, Ferra C, Garnier F, Loiseau P, Garcia J, Lecchi L, Kogler G, Beguin Y, Navarrete C, Devos T, Ionescu I, Boudjedir K, Herr AL, Gluckman E, Rocha V; Eurocord-Netcord and Acute Leukaemia Working Party of the EBMT. KIR-ligand incompatibility in the graft-versus-host direction improves outcomes after umbilical cord blood transplantation for acute leukemia. Leukemia. 2009 Mar;23(3):492-500. doi: 10.1038/leu.2008.365. Epub 2009 Jan 8. PMID 19151783
- [Background] Merindol N, Charrier E, Duval M, Soudeyns H. Complementary and contrasting roles of NK cells and T cells in pediatric umbilical cord blood transplantation. J Leukoc Biol. 2011 Jul;90(1):49-60. doi: 10.1189/jlb.0111007. Epub 2011 Mar 2. PMID 21367975
- [Background] Delaney C, Heimfeld S, Brashem-Stein C, Voorhies H, Manger RL, Bernstein ID. Notch-mediated expansion of human cord blood progenitor cells capable of rapid myeloid reconstitution. Nat Med. 2010 Feb;16(2):232-6. doi: 10.1038/nm.2080. Epub 2010 Jan 17. PMID 20081862
- [Background] Shpall EJ, Bollard CM, Brunstein C. Novel cord blood transplant therapies. Biol Blood Marrow Transplant. 2011 Jan;17(1 Suppl):S39-45. doi: 10.1016/j.bbmt.2010.10.004. Epub 2010 Oct 15. No abstract available. PMID 20951821
- [Background] Bautista G, Cabrera JR, Regidor C, Fores R, Garcia-Marco JA, Ojeda E, Sanjuan I, Ruiz E, Krsnik I, Navarro B, Gil S, Magro E, de Laiglesia A, Gonzalo-Daganzo R, Martin-Donaire T, Rico M, Millan I, Fernandez MN. Cord blood transplants supported by co-infusion of mobilized hematopoietic stem cells from a third-party donor. Bone Marrow Transplant. 2009 Mar;43(5):365-73. doi: 10.1038/bmt.2008.329. Epub 2008 Oct 13. PMID 18850019
- [Background] Liu H, Rich ES, Godley L, Odenike O, Joseph L, Marino S, Kline J, Nguyen V, Cunningham J, Larson RA, del Cerro P, Schroeder L, Pape L, Stock W, Wickrema A, Artz AS, van Besien K. Reduced-intensity conditioning with combined haploidentical and cord blood transplantation results in rapid engraftment, low GVHD, and durable remissions. Blood. 2011 Dec 8;118(24):6438-45. doi: 10.1182/blood-2011-08-372508. Epub 2011 Oct 5. PMID 21976674
- [Background] Eapen M, Klein JP, Sanz GF, Spellman S, Ruggeri A, Anasetti C, Brown M, Champlin RE, Garcia-Lopez J, Hattersely G, Koegler G, Laughlin MJ, Michel G, Nabhan SK, Smith FO, Horowitz MM, Gluckman E, Rocha V; Eurocord-European Group for Blood and Marrow Transplantation; Netcord; Center for International Blood and Marrow Transplant Research. Effect of donor-recipient HLA matching at HLA A, B, C, and DRB1 on outcomes after umbilical-cord blood transplantation for leukaemia and myelodysplastic syndrome: a retrospective analysis. Lancet Oncol. 2011 Dec;12(13):1214-21. doi: 10.1016/S1470-2045(11)70260-1. Epub 2011 Oct 6. PMID 21982422
- [Background] Ponce DM, Zheng J, Gonzales AM, Lubin M, Heller G, Castro-Malaspina H, Giralt S, Hsu K, Jakubowski AA, Jenq RR, Koehne G, Papadopoulos EB, Perales MA, van den Brink MR, Young JW, Boulad F, Kernan NA, Kobos R, Prockop S, Scaradavou A, Small T, O'Reilly RJ, Barker JN. Reduced late mortality risk contributes to similar survival after double-unit cord blood transplantation compared with related and unrelated donor hematopoietic stem cell transplantation. Biol Blood Marrow Transplant. 2011 Sep;17(9):1316-26. doi: 10.1016/j.bbmt.2011.01.006. Epub 2011 Jan 11. PMID 21232625
- [Background] Scaradavou A, Smith KM, Hawke R, Schaible A, Abboud M, Kernan NA, Young JW, Barker JN. Cord blood units with low CD34+ cell viability have a low probability of engraftment after double unit transplantation. Biol Blood Marrow Transplant. 2010 Apr;16(4):500-8. doi: 10.1016/j.bbmt.2009.11.013. Epub 2009 Nov 22. PMID 19932758
- [Background] Takanashi M, Atsuta Y, Fujiwara K, Kodo H, Kai S, Sato H, Kohsaki M, Azuma H, Tanaka H, Ogawa A, Nakajima K, Kato S. The impact of anti-HLA antibodies on unrelated cord blood transplantations. Blood. 2010 Oct 14;116(15):2839-46. doi: 10.1182/blood-2009-10-249219. Epub 2010 Jul 13. PMID 20628152
- [Background] Cutler C, Kim HT, Sun L, Sese D, Glotzbecker B, Armand P, Koreth J, Ho V, Alyea E, Ballen K, Ritz J, Soiffer RJ, Milford E, Antin JH. Donor-specific anti-HLA antibodies predict outcome in double umbilical cord blood transplantation. Blood. 2011 Dec 15;118(25):6691-7. doi: 10.1182/blood-2011-05-355263. Epub 2011 Sep 22. PMID 21940825
- [Background] Brunstein CG, Noreen H, DeFor TE, Maurer D, Miller JS, Wagner JE. Anti-HLA antibodies in double umbilical cord blood transplantation. Biol Blood Marrow Transplant. 2011 Nov;17(11):1704-8. doi: 10.1016/j.bbmt.2011.04.013. Epub 2011 May 3. PMID 21601639
- [Background] van Rood JJ, Stevens CE, Smits J, Carrier C, Carpenter C, Scaradavou A. Reexposure of cord blood to noninherited maternal HLA antigens improves transplant outcome in hematological malignancies. Proc Natl Acad Sci U S A. 2009 Nov 24;106(47):19952-7. doi: 10.1073/pnas.0910310106. Epub 2009 Nov 9. PMID 19901324
- [Background] van Rood JJ, Scaradavou A, Stevens CE. Indirect evidence that maternal microchimerism in cord blood mediates a graft-versus-leukemia effect in cord blood transplantation. Proc Natl Acad Sci U S A. 2012 Feb 14;109(7):2509-14. doi: 10.1073/pnas.1119541109. Epub 2012 Jan 9. PMID 22232664
- [Background] Stern M, de Angelis C, Urbani E, Mancusi A, Aversa F, Velardi A, Ruggeri L. Natural killer-cell KIR repertoire reconstitution after haploidentical SCT. Bone Marrow Transplant. 2010 Nov;45(11):1607-10. doi: 10.1038/bmt.2010.19. Epub 2010 Feb 22. PMID 20173785
- [Background] Ballen KK, Barker JN. Has umbilical cord blood transplantation for AML become mainstream? Curr Opin Hematol. 2013 Mar;20(2):144-9. doi: 10.1097/MOH.0b013e32835dd936. PMID 23314845
- See also: Blood and Tissue Bank of Catalonia — http://www.bancsang.net
- See also: Hospital de Sant Pau — http://www.santpau.es
- See also: Hospital Vall d'Hebron — http://www.vhebron.net
- See also: Hospital Universitari de Bellvitge — http://www.bellvitgehospital.cat
- See also: Hospital Universitari Germans Trias i Pujol — http://www.gencat.cat/ics/germanstrias
- See also: Institut Hospital del Mar d'Investigacions Mèdiques — http://www.imim.cat